CLINICAL TRIAL: NCT03375619
Title: Long-term Follow-up Study of Patients Receiving CAR-T Cells
Status: Recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Nirav Shah, Associate Professor, Medical College of Wisconsin
Other Study IDs: PRO30317
Record Dates: First submitted 2017-12-07; First posted 2017-12-18 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukemia; Lymphomas Non-Hodgkin's B-Cell; Lymphoma, Small Lymphocytic; Mantle Cell Lymphoma; Central Nervous System Lymphoma; Diffuse Large B Cell Lymphoma; Follicular Lymphoma; Burkitt Lymphoma; Multiple Myeloma
Keywords: CAR-T Cell Therapy; chimeric antigen receptor
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Burkitt Lymphoma; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants who received CAR-T cells.: Participants who received CAR-T cells at Froedtert Hospital & the Medical College of Wisconsin in clinical trials (e.g., NCT05976555, NCT05094206, NCT05990465, NCT03019055 or NCT04186520).
  Interventions: Other: Long-Term Follow-Up of Participants who Received CAR-T cells

INTERVENTIONS:
Other: Long-Term Follow-Up of Participants who Received CAR-T cells — No study drug is administered in this study. Participants who received CAR-T cells in a previous trial will be evaluated in this trial for long-term safety and efficacy.

SUMMARY:
This protocol is designed as a long-term follow-up study of participants who will receive CAR-T cells as part of a clinical trial at the Medical College of Wisconsin/ Froedtert Hospital. The clinical trials include the following:

Phase 1 Study of CAR-20/19-T Cells in Patients with Relapsed Refractory B Cell Malignancies (NCT03019055); Phase I Trial of BCMA-TGF-BETA CAR-T Cells in Relapsed, Refractory Myeloma (NCT05976555); CAR20.19.22 T-cells in Relapsed, Refractory B-cell Malignancies (NCT05094206); LV20.19 CAR T-Cells in Combination With Pirtobrutinib for Relapsed, Refractory B-cell Malignancies (NCT05990465); CAR-20/19-T Cells in Patients With Relapsed Refractory B Cell Malignancies (NCT04186520)

DETAILED DESCRIPTION:
The objective is to follow participants receiving CAR-T cells from years 2 to 15 post-treatment for persistence of CAR-T cells, development of secondary malignancies, or other medical complications.

ELIGIBILITY:
Inclusion Criteria:

* All participants who enrolled in a CAR-T study at Froedtert Hospital & the Medical College of Wisconsin.

Exclusion Criteria:

* There are no exclusion criteria for this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants who enrolled in a CAR-T study at Froedtert Hospital & the Medical College of Wisconsin.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2035-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the incidence of a new malignancy at 5 years. | Baseline to five years.
  The number of subjects with new malignancy.
Change from baseline in the incidence of a new malignancy at 10 years. | Baseline to 10 years.
  The number of subjects with new malignancy.
Change from baseline in the incidence of a new malignancy at 15 years. | Baseline to 15 years.
  The number of subjects with new malignancy.

CONTACTS AND LOCATIONS:
Overall Officials: Nirav Shah, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No